CLINICAL TRIAL: NCT03479957
Title: Remotely Monitored and Coached Exercise Based Cardiac Rehabilitation in Northern Sweden l
Brief Title: Remotely Monitored and Coached Cardiac Rehabilitation Northern Sweden
Acronym: RECREATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Camilla Sandberg, Principal Investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RemoteCR SWE
Record Dates: First submitted 2018-03-15; First posted 2018-03-27 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMOTE-CR (Experimental): Remotely monitored and coached exercise training in real time using the REMOTE-CR system. The patients randomized to remotely monitored exercise can either work out with self-selected activities e.g. Nordic-walking, cycling, skiing or participate in supervised exercise session via video link.
  Interventions: Behavioral: REMOTE-CR
- Usual care (Other): The patients randomized to be controls will receive individualized information and instructions regarding current exercise recommendations but will not be monitored or coached during their exercise sessions (usual care).
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: REMOTE-CR — The patients randomized to remotely monitored exercise can either work out with self-selected activities e.g. Nordic-walking, cycling, skiing or participate in supervised exercise session via video link. Remotely monitored exercise training sessions will be offered monday-friday 13.00-16.00.
  Arms: REMOTE-CR
Other: Control — The patients randomized to be controls will receive individualized information and instructions regarding current exercise recommendations but will not be monitored or coached during their exercise sessions (usual care)
  Arms: Usual care

SUMMARY:
Supervised exercise is an essential component of contemporary center-based cardiac rehabilitation (CR) programs. Despite the proven effectiveness, uptake and adherence to supervised exercise-based CR (exCR) remains suboptimal (approximately 50%), especially in rural and remote areas of Sweden. The main reasons for low participation rate in centre-based exCR are different accessibility barriers i.e. long distances, transportation problems or employment commitments. In this randomised clinical trial, the overall aim is to evaluate the effectiveness of, home-based, remotely monitored and coached exCR using the REMOTE-CR system compared to home-based exCR based on individualized information regarding current exercise recommendations but without monitoring and coaching (usual care) to improve exercise capacity. Our hypothesis is that remotely monitored and coached exCR will improve exercise capacity to a greater extent than home-based exCR without monitoring and coaching (usual care).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled appointment with physiotherapist for follow-up after cardiac event: ----Myocardial Infarction (MI)
* Per cutaneous coronary intervention (PCI) due to MI or angina pectoris
* Open heart surgery due to coronary artery disease or valvar disease
* Living in the catchment area of Heart centre, University Hospital of Umeå.

Exclusion Criteria:

* Clinically unstable
* Postoperative infection
* Comorbidity affecting ability to participate in exCR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-02-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in submaximal aerobic exercise capacity | Baseline and 12 weeks
  The aerobic exercise capacity (W) will be evaluated using a standardised submaximal exercise test on cycle ergometer

SECONDARY OUTCOMES:
Muscle endurance capacity | Baseline and 12 weeks
  Number of repetitions achieved during test of Unilateral isotonic shoulder flexion and Unilateral isotonic heel-lift
Isometric grip strength | Baseline and 12 weeks
  Isometric grip strength will be evaluated using a hydraulic hand dynamometer
Self-reported physical activity using theInternational Physical Activity Questionnaire | Baseline and 12 weeks
  International Physical Activity Questionnaire: Results will be presented as a continuous variable, total metabolic equivalent (MET) minutes per week, where a higher score indicates a higher physical activity level. Result will also be presented as a categorical variable:
  High Physical activity level: achieving a total physical activity of at least 3000 MET-minutes/week.
  Moderate physical activity: achieving a minimum of at least 600 MET-minutes per week.
  Low physical activity level: not achieving the minimum of 600 MET minutes per week
Self-reported physical activity using the physical activity scale br Frändin and Grimby | Baseline and 12 weeks
  The Activity scale by Frändin and Grimby describes 6 levels of physical activity. The scale includes 6 items that ranges from 1 indicating mostly physically inactive to 6 indicating a very high physical activity level.
Kinesiophobia (fear of movement) | Baseline and 12 weeks
  The Swedish version of the Tampa scale for Kinesiophobia Heart (TSK-SV Heart) The scale comprises 17 items assessing subjective rating of kinesiophobia. The total score varies between 17-68 and a score >37 defines a high level of kinesofobia.

OTHER OUTCOMES:
Evaluation of change the participation rate in supervised cardiac rehabilitation | 12 weeks
  Evaluation of change the participation rate can be enhanced using the REMOTE -CR system
Patients experiences of REMOTE-CR and and exercise led via video link | 12 weeks
  The study participants experience of the REMOTE-CR system and exercise sessions via video link will be evaluated using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Sandberg, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No